CLINICAL TRIAL: NCT06919042
Title: A Prospective Single-center Study for Evaluation of the Effectiveness of Pulsed Acoustic Cellular Expression Technology on Post-Operative Soft Tissue Fibrosis.
Brief Title: Shockwave in Postoperative Breast Reconstruction Fibrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Robert Galiano, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00221726
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Fibrosis Breast
Keywords: breast fibrosis; postoperative fibrosis; shockwave therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (No Intervention): The control arm receives eight sessions of a sham (placebo) version of the therapy.
- Intervention (Experimental): The intervention arm receives eight sessions of Pulsed Acoustic Cellular Expression (PACE) therapy delivered twice weekly for four weeks at level E2
  Interventions: Device: Pulsed Acoustic Cellular Expression therapy

INTERVENTIONS:
Device: Pulsed Acoustic Cellular Expression therapy — The therapy involves the delivery of targeted acoustic energy that initiates cellular mechanotransduction pathways, inducing beneficial biological responses such as enhanced angiogenesis, modulation of fibroblast proliferation and differentiation, and reorganization of aberrant extracellular matrix components.
  Arms: Intervention

SUMMARY:
This study evaluates the potential for extracorporeal shockwave therapy to reduce post-operative soft tissue fibrosis.

DETAILED DESCRIPTION:
This study was conducted as a single-blind, randomized controlled trial (RCT) to evaluate the efficacy of acoustic shockwave therapy in treating post-surgical fibrosis following breast reconstruction. The intervention period spanned four weeks, during which participants received a total of eight treatment sessions-two sessions per week. Participants returned for follow-up evaluation at three months. Patients were randomized to either the intervention arm, which received active shockwave therapy, or the control arm, which received a sham (placebo) version of the therapy. Randomization was performed using a computer. Participants were blinded to treatment group allocation; however, clinicians administering the therapy were not, due to the procedural nature of the intervention.

Eligible patients included adult females with clinically diagnosed postoperative fibrosis after breast reconstruction. Patients with prior radiation exposure or capsular contracture were included and stratified by indication into three categories: post-breast reconstruction fibrosis without radiation, (1) post-breast reconstruction fibrosis following radiation, and (2) post-breast reconstruction fibrosis with capsular contracture. Demographic data including age and race/ethnicity were collected. Patients with active infection, systemic illness, or pregnancy were excluded.

The shockwave therapy group received eight sessions of Pulsed Acoustic Cellular Expression (PACE) therapy delivered twice weekly for four weeks at level E2. Therapy parameters (e.g. number of pulses) were adjusted based on the anatomical location and severity of fibrosis, in accordance with manufacturer guidelines. The control group underwent the same schedule and treatment setup using the same equipment, but with the shockwave component disabled to serve as a placebo.

Outcome measures were assessed at each session (1-8) and at 3 months. Patient-reported outcomes included perceived change in fibrosis size (rated 1-10, with 10 being the greatest reduction), softness/pliability (10 being softest), pain (10 indicating worst pain), and shoulder mobility (10 indicating greatest mobility). Observer-based clinical outcomes included assessments of size (10 = largest), contour (10 = worst), firmness (10 = hardest), shoulder mobility (10=full mobility) and overall impression (10 = worst quality). In addition, scar area was measured objectively in square millimeters using caliper measurements. Video recordings of the treated areas were collected at visit to qualitatively assess visual changes over time. In addition to clinical and patient-reported outcomes, point-of-care handheld ultrasound (POCUS) was used to qualitatively assess tissue characteristics at baseline and at session 8 follow-up. Ultrasound evaluations were performed using a standardized protocol by a trained study team member. Recordings were analyzed qualitatively using a 5-point Likert scale across five domains: (1) fibrosis size, (2) echogenicity, (3) homogeneity, and (4) boundary definition. Higher scores indicated more favorable healing outcomes. Comparisons between treatment and placebo groups were conducted using the Wilcoxon rank-sum test due to the ordinal nature of the scoring system.

ELIGIBILITY:
Inclusion Criteria:

* Subjects greater than 18 years of age.
* Subjects who have undergone plastic surgery procedures and present in the post-operative period with soft tissue firmness suggestive of subcutaneous/parenchymal fibrosis.

Exclusion Criteria:

* Subjects with cardiac pacemakers
* Other medical or psychiatric condition that may increase the risk associated with study participation, may complicate subject compliance, or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
* Proximity of fibrotic tissue directly adjacent to bone
* Face/neck areas are excluded
* Patients who, in the opinion of the investigator, would not be compliant with the schedule of study visits

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Subcutaneous Fibrosis Mass | One month
  Reduction in size of subcutaneous fibrosis mass assess clinically by PI, point-of-care ultrasound, caliper measurements, and objective/subjective measures by an observer and the patient.

SECONDARY OUTCOMES:
Pain Score | One month
  Pain scores and reduction
Adverse Events | Three months
  Any adverse events associated with the focused shockwave therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Lavin Pavilion Suite 2060, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen AT, Chon J, Li RA, Melnick BA, Abu-Romman A, Laiwalla R, Adam TH, Galiano RD. Extracorporeal shockwave therapy improves post-breast reconstruction fibrosis: A randomized controlled blinded clinical trial. J Plast Reconstr Aesthet Surg. 2025 Nov;110:7-17. doi: 10.1016/j.bjps.2025.08.045. Epub 2025 Sep 9. PMID 41038043